CLINICAL TRIAL: NCT04308668
Title: Post-exposure Prophylaxis or Preemptive Therapy for SARS-Coronavirus-2: A Pragmatic Randomized Clinical Trial
Brief Title: Post-exposure Prophylaxis / Preemptive Therapy for SARS-Coronavirus-2
Acronym: COVID-19 PEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); University of Manitoba (Other); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MED-2020-28673
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Corona Virus Infection; Acute Respiratory Distress Syndrome; SARS-CoV Infection; Coronavirus; Coronavirus Infections
Keywords: COVID-19; Corona Virus; SARS-COV-2; Coronavirus
MeSH Terms: conditions — Coronavirus Infections; Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome; COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Asymptomatic participants are randomized and analyzed separate from symptomatic participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants in this arm will receive the study drug.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — 200mg tablet; 800 mg orally once, followed in 6 to 8 hours by 600 mg, then 600mg once a day for 4 consecutive days
  Other Names: Plaquenil
  Arms: Treatment
Other: Placebo — 4 placebo tablets once, followed in 6 to 8 hours by 3 tablets, then 3 tablets once-a-day for 4 consecutive days
  Arms: Placebo

SUMMARY:
Study Objective:

1. To test if post-exposure prophylaxis with hydroxychloroquine can prevent symptomatic COVID-19 disease after known exposure to the SARS-CoV-2 coronavirus.
2. To test if early preemptive hydroxychloroquine therapy can prevent disease progression in persons with known symptomatic COVID-19 disease, decreasing hospitalizations and symptom severity.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a rapidly emerging viral infection causing COVID19. The current strategy uses a public health model of identifying infected cases, isolation, and quarantine to stop transmission. Once exposed, observation is standard-of-care. Therapy is generally not given to persons who are not hospitalized. The doses of hydroxychloroquine being used are within the normal standard FDA-approved doses.

Hydroxychloroquine may have antiviral effects against SARS-COV2 which may prevent COVID-19 disease or early preemptive therapy may decrease disease severity. This trial will use a modification of standard malaria dosing of hydroxychloroquine to provide post-exposure prophylaxis to prevent disease or preemptive therapy for those with early symptoms. People around the the United States and Canada can participate to help answer this critically important question. No in-person visits are needed.

This trial is targeting 5 groups of people NATIONWIDE to participate:

1. If you are symptomatic with a positive COVID-19 test within the first 4 days of symptoms and are not hospitalized; OR
2. If you live with someone who has been diagnosed with COVID-19, with your last exposure within the last 4 days, and do not have any symptoms; OR
3. If you live with someone who has been diagnosed with COVID-19, and your symptoms started within the last 4 days; OR
4. If you have had occupational exposure with known exposure to someone with lab-confirmed COVID-19 within the last 4 days and do not have symptoms; OR
5. If you have had occupational exposure with known exposure to someone with lab-confirmed COVID-19 within the last 4 days AND have compatible symptoms starting within the last 4 days;

You may participate if you live anywhere in the United States (including territories) or in the Canadian Provinces of Quebec, Manitoba, Alberta, or Ontario.

For information on how to participate in the research trial, go to covidpep.umn.edu or email covid19@umn.edu for instructions. Please check your spam folder if you email.

In Canada, for trial information, please go to: www.covid-19research.ca

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Exposure to a COVID19 case within 4 days as either a household contact or occupational exposure, OR
* Symptomatic COVID19 case with confirmed diagnosis within 4 days of symptom onset OR symptomatic high risk exposure with known COVID19 contact and within 4 days of symptom onset;

Exclusion Criteria:

* Current hospitalization
* Allergy to hydroxychloroquine
* Retinal eye disease
* Known glucose-6 phosphate dehydrogenase (G-6-PD) deficiency
* Known chronic kidney disease, stage 4 or 5 or receiving dialysis
* Structural or ischemic heart disease
* Personal or Family History of Prolonged QT syndrome
* Weight < 50 kg
* Known Porphyria
* Current use of: hydroxychloroquine or cardiac medicines of: flecainide, Tambocor; amiodarone, Cordarone, Pacerone; digoxin or Digox, Digitek, Lanoxin; procainamide or Procan, Procanbid, propafenone, Rythmal, sotalol;
* Current use of medicines which prolong the QT interval including:

  * Antimicrobials: levofloxacin, ciprofloxacin, moxifloxacin, azithromycin, clarithromycin, erythromycin, ketoconazole, itraconazole, or mefloquine
  * Antidepressants: amitriptyline, citalopram, desipramine, escitalopram, imipramine, doxepin, fluoxetine, wellbutrin, or venlafaxine
  * Antipsychotic or mood stabilizers: haloperidol, droperidol, lithium, quetiapine, thioridazine, ziprasidone
  * Methadone
  * Sumatriptan, zolmitriptan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1312 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Boulware, MD, MPH, Principal Investigator — University of Minnesota
Locations (5):
- United States (2):
  - Nationwide Enrollment via Internet, please email: covid19@umn.edu, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - Research Institute of the McGill University Heath Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
De-identified dataset will be available within 1 month of publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: at time of publication
Access Criteria: To be publicly provided. Please register at the website to receive the dataset.
URL: https://covidpep.umn.edu/data

REFERENCES:
- [Background] Lother SA, Abassi M, Agostinis A, Bangdiwala AS, Cheng MP, Drobot G, Engen N, Hullsiek KH, Kelly LE, Lee TC, Lofgren SM, MacKenzie LJ, Marten N, McDonald EG, Okafor EC, Pastick KA, Pullen MF, Rajasingham R, Schwartz I, Skipper CP, Turgeon AF, Zarychanski R, Boulware DR. Post-exposure prophylaxis or pre-emptive therapy for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2): study protocol for a pragmatic randomized-controlled trial. Can J Anaesth. 2020 Sep;67(9):1201-1211. doi: 10.1007/s12630-020-01684-7. Epub 2020 May 7. PMID 32383125
- [Background] Pastick KA, Okafor EC, Wang F, Lofgren SM, Skipper CP, Nicol MR, Pullen MF, Rajasingham R, McDonald EG, Lee TC, Schwartz IS, Kelly LE, Lother SA, Mitja O, Letang E, Abassi M, Boulware DR. Review: Hydroxychloroquine and Chloroquine for Treatment of SARS-CoV-2 (COVID-19). Open Forum Infect Dis. 2020 Apr 15;7(4):ofaa130. doi: 10.1093/ofid/ofaa130. eCollection 2020 Apr. PMID 32363212
- [Background] Al-Kofahi M, Jacobson P, Boulware DR, Matas A, Kandaswamy R, Jaber MM, Rajasingham R, Young JH, Nicol MR. Finding the Dose for Hydroxychloroquine Prophylaxis for COVID-19: The Desperate Search for Effectiveness. Clin Pharmacol Ther. 2020 Oct;108(4):766-769. doi: 10.1002/cpt.1874. Epub 2020 Jun 1. PMID 32344449
- [Background] Ingraham NE, Boulware D, Sparks MA, Schacker T, Benson B, Sparks JA, Murray T, Connett J, Chipman JG, Charles A, Tignanelli CJ. Shining a light on the evidence for hydroxychloroquine in SARS-CoV-2. Crit Care. 2020 Apr 28;24(1):182. doi: 10.1186/s13054-020-02894-7. No abstract available. PMID 32345336
- [Background] Pullen MF, Pastick KA, Williams DA, Nascene AA, Bangdiwala AS, Okafor EC, Hullsiek KH, Skipper CP, Lofgren SM, Engen N, Abassi M, McDonald EG, Lee TC, Rajasingham R, Boulware DR. Lessons Learned From Conducting Internet-Based Randomized Clinical Trials During a Global Pandemic. Open Forum Infect Dis. 2020 Dec 28;8(2):ofaa602. doi: 10.1093/ofid/ofaa602. eCollection 2021 Feb. PMID 33553471
- [Background] Okafor EC, Pastick KA, Rajasingham R. Hydroxychloroquine as Postexposure Prophylaxis for Covid-19. Reply. N Engl J Med. 2020 Sep 10;383(11):1089. doi: 10.1056/NEJMc2023617. Epub 2020 Jul 15. No abstract available. PMID 32668109
- [Result] Boulware DR, Pullen MF, Bangdiwala AS, Pastick KA, Lofgren SM, Okafor EC, Skipper CP, Nascene AA, Nicol MR, Abassi M, Engen NW, Cheng MP, LaBar D, Lother SA, MacKenzie LJ, Drobot G, Marten N, Zarychanski R, Kelly LE, Schwartz IS, McDonald EG, Rajasingham R, Lee TC, Hullsiek KH. A Randomized Trial of Hydroxychloroquine as Postexposure Prophylaxis for Covid-19. N Engl J Med. 2020 Aug 6;383(6):517-525. doi: 10.1056/NEJMoa2016638. Epub 2020 Jun 3. PMID 32492293
- [Result] Skipper CP, Pastick KA, Engen NW, Bangdiwala AS, Abassi M, Lofgren SM, Williams DA, Okafor EC, Pullen MF, Nicol MR, Nascene AA, Hullsiek KH, Cheng MP, Luke D, Lother SA, MacKenzie LJ, Drobot G, Kelly LE, Schwartz IS, Zarychanski R, McDonald EG, Lee TC, Rajasingham R, Boulware DR. Hydroxychloroquine in Nonhospitalized Adults With Early COVID-19 : A Randomized Trial. Ann Intern Med. 2020 Oct 20;173(8):623-631. doi: 10.7326/M20-4207. Epub 2020 Jul 16. PMID 32673060
- [Result] Lofgren SM, Nicol MR, Bangdiwala AS, Pastick KA, Okafor EC, Skipper CP, Pullen MF, Engen NW, Abassi M, Williams DA, Nascene AA, Axelrod ML, Lother SA, MacKenzie LJ, Drobot G, Marten N, Cheng MP, Zarychanski R, Schwartz IS, Silverman M, Chagla Z, Kelly LE, McDonald EG, Lee TC, Hullsiek KH, Boulware DR, Rajasingham R. Safety of Hydroxychloroquine Among Outpatient Clinical Trial Participants for COVID-19. Open Forum Infect Dis. 2020 Oct 19;7(11):ofaa500. doi: 10.1093/ofid/ofaa500. eCollection 2020 Nov. PMID 33204764
- [Result] Skipper CP, Boulware DR. Hydroxychloroquine in Nonhospitalized Adults With Early COVID-19. Ann Intern Med. 2021 Mar;174(3):434-435. doi: 10.7326/L20-1426. No abstract available. PMID 33721539
- [Result] Nicol MR, Boulware DR, Rajasingham R. Reply to Neves. Clin Infect Dis. 2021 Oct 5;73(7):e1772-e1774. doi: 10.1093/cid/ciaa1809. No abstract available. PMID 33274360
- [Derived] Akhtar S, Das JK, Ismail T, Wahid M, Saeed W, Bhutta ZA. Nutritional perspectives for the prevention and mitigation of COVID-19. Nutr Rev. 2021 Feb 11;79(3):289-300. doi: 10.1093/nutrit/nuaa063. PMID 33570583
- Available data/document: Individual Participant Data Set — http://www.covidpep.umn.edu/data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 658 | 654
Completed | 622 | 612
Not Completed | 36 | 42
Not completed — Lost to Follow-up | 32 | 38
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 658 | 654 | 1312
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12) | 42 (12) | 42 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: While biological sex at birth was the question, 4 persons in each arm did not identify as male or female.
  Participants
    Sex: number analyzed (Participants) | 654 | 650 | 1304
    Sex: Female | 354 | 336 | 690
    Sex: Male | 300 | 314 | 614
    Non-binary: number analyzed (Participants) | 4 | 4 | 8
    Non-binary: Female | 2 | 2 | 4
    Non-binary: Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants could identify as more than one Race/Ethnicity
  Participants
    American Indian or Alaska Native | 4 | 2 | 6
    Asian/South Asian | 204 | 206 | 410
    Native Hawaiian or Pacific Islander | 5 | 4 | 9
    Black or African American | 28 | 24 | 52
    White | 363 | 379 | 742
    Hispanic or Latino | 37 | 36 | 73
    Middle Eastern | 14 | 9 | 23
    Unknown/Not Reported | 12 | 10 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 30 | 29 | 59
  United States | 628 | 625 | 1253

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Active COVID-19 Disease at Day 14 Among Those Who Were Asymptomatic at Baseline
Description: Number of participants at 14 days post enrollment with active COVID19 disease among those who were asymptomatic at baseline.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 414 | 407
Participants | 49 | 58
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.35, Fisher Exact; Mean Difference (Net) = -2.4, 95% CI 2-sided [-7.0 to 2.2] — Values represent percentages. Experimental treatment arm compared with the placebo control arm

2. Primary Outcome: Change in Disease Severity Over 14 Days Among Those Who Are Symptomatic at Baseline
Description: Visual Analog Scale 0-10 score of rating overall symptom severity (0 = no symptoms; 10 = most severe)
Time Frame: baseline and 14 days
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 212 | 211
score on a scale | -2.6 (.12) | -2.33 (.12)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.117, Mixed Models Analysis; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.61 to 0.27]

3. Secondary Outcome: Rate of Hospitalization
Description: Outcome reported as the number of participants in each arm who require hospitalization for COVID19-related disease.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 645 | 641
Participants | 5 | 9

4. Secondary Outcome: Rate of Death
Description: Outcome reported as the number of participants in each arm who expire due to COVID-19-related disease through study completion of 14 days. For those hospitalized within the 14-day study period, the protocol specified follow up would occur for up to 90 days to capture the final outcome of participants' hospitalization. Approximately 30-days was the maximal follow up for hospitalization outcome needed in the trial.
Time Frame: Approximately 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 645 | 641
Participants | 1 | 1

5. Secondary Outcome: Rate of Confirmed SARS-CoV-2 Detection
Description: Outcome reported as the number of participants in each arm who have confirmed SARS-CoV-2 infection.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 414 | 407
Participants | 11 | 9

6. Secondary Outcome: Occurrence of Symptoms Compatible With COVID-19 (Possible Disease)
Description: Outcome reported as the number of participants in each arm who self-report symptoms compatible with COVID-19 infection.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 414 | 407
Participants | 48 | 55

7. Secondary Outcome: Rate of All-Cause Study Medicine Discontinuation or Withdrawal
Description: Outcome reported as the number of participants in each arm who discontinue or withdraw medication use for any reason.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 645 | 641
Participants | 97 | 63

8. Secondary Outcome: Overall Symptom Severity at 5 and 14 Days
Description: Visual Analog Scale 0-10 score of rating overall symptom severity (0 = no symptoms; 10 = most severe)
Time Frame: 5 and 14 days
Population: Early preemptive treatment trial (n=423 symptomatic participants with data)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 212 | 211
score on a scale
  Day 5 | -2.22 [-2.53 to -1.9] | -2.05 [-2.37 to -1.73]
  Day 14 | -3.36 [-3.62 to -3.09] | -3.08 [-3.35 to -2.81]

9. Secondary Outcome: Number of Participants With Severe COVID-19 Disease at 14 Days Among Those Who Are Symptomatic at Trial Entry
Description: Participants will self-report disease severity status as one of the following 3 options; no COVID19 illness (score of 1), COVID19 illness with no hospitalization (score of 2), or COVID19 illness with hospitalization or death (score of 3). Increased scale score indicates greater disease severity. Outcome is reported as the number of participants who report a score of 3.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 231 | 234
Participants | 5 | 8

ADVERSE EVENTS:
Time Frame: Approximately 30-days
Description: Reporting period was for onset of adverse events within 14 days. All hospitalizations were followed for up to 90 days for final resolution of outcome. Approximately 30 days was the maximal duration needed to capture final outcome.
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 1/658 | 1/654
Serious Adverse Events (participants affected / at risk) | 6/658 | 11/654
Other Adverse Events (participants affected / at risk) | 367/658 | 148/654
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=658) | Placebo (N=654)
COVID-related hospitalization (Infections and infestations) | 6 (6) | 9 (9) — n=5 vs. n=8 hospitalizations in early treatment population, n=1 vs. n=1 hospitalizations in postexposure prophylaxis population
Hospitalizations not related to COVID or study medicine (Cardiac disorders) | 0 (0) | 2 (2) — Adjudication was conducted by blinded investigators.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=658) | Placebo (N=654)
Nausea or upset stomach (Gastrointestinal disorders) | 146 (146) | 53 (53)
Diarrhea, abdominal pain, vomiting (Gastrointestinal disorders) | 131 (131) | 35 (35)
Irritability, dizziness, vertigo (General disorders) | 39 (39) | 26 (26)
Tinnitus (Ear and labyrinth disorders) | 16 (16) | 8 (8)
Headache (General disorders) | 15 (15) | 8 (8)
Visual changes (Eye disorders) | 7 (7) | 5 (5)
Skin reaction (Skin and subcutaneous tissue disorders) | 10 (10) | 4 (4)
Taste change or dry mouth (General disorders) | 3 (3) | 3 (3)
Allergic reaction (non-anaphylaxis) (Immune system disorders) | 6 (6) | 1 (1)
Hot flashes, night sweats, palpitations (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Panic (Psychiatric disorders) | 0 (0) | 1 (1)
Other (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04308668/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04308668/ICF_001.pdf